CLINICAL TRIAL: NCT04308941
Title: Tonometry Precision and Accuracy During PROSE Scleral Lens Wear: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Sight (Other)
Responsible Party: Principal Investigator, Daniel C Brocks, Principal Invesigator, Boston Sight
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: BFS-KR-IOP-02
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Intraocular Pressure and PROSE Lens
MeSH Terms: interventions — Intraocular Pressure

STUDY DESIGN:
Intervention Model Description: The first 10 subjects will be randomly chosen for the first cohort (scleral TonoPen), the second 10 subjects will be randomly chosen for the second cohort (scleral pneumatonometry), and the third 10 subjects will be randomly chosen for the third cohort (Diaton).
Masking Description: Subjects will be enrolled in each cohort sequentially there is no masking of procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Scleral Tonopen (Active Comparator): The first 10 subjects will be randomly chosen for the first cohort (scleral TonoPen)
  Interventions: Diagnostic Test: Intraocular pressure
- Scleral Pneumatonometer (Active Comparator): The second 10 subjects will be randomly chosen for the second cohort (scleral pneumatonometry)
  Interventions: Diagnostic Test: Intraocular pressure
- Diaton (Active Comparator): The third 10 subjects will be randomly chosen for the third cohort (Diaton).
  Interventions: Diagnostic Test: Intraocular pressure

INTERVENTIONS:
Diagnostic Test: Intraocular pressure — The intraocular pressure will be measured using one of three devices

SUMMARY:
The goal of this research is to determine the reproducibility of measurements of intraocular pressure (IOP) when a scleral lens is on the eye. The PROSE device (PD) is a specialized scleral lens that is filled with preservative-free saline and then applied to the eye in order to treat a variety of ocular conditions. The fit of the PROSE device is optimized to land gently on the conjunctival tissue overlying the sclera while completely vaulting the cornea and limbus without touch.

Because the PROSE device vaults and therefore covers the cornea, measuring IOP during PROSE wear is challenging as traditional techniques rely on corneal contact (i.e. Goldmann tonometry, iCare, pneumatonometry, etc.). Measuring IOP before insertion and after removal of the PROSE device likely does not correspond to the true IOP when the PROSE device is actively on the eye.

This is a prospective study of the reproducibility of three non-traditional means of IOP measurements: scleral tonopen, scleral pneumatonometry, and transpalpebral Diaton tonometer. Evaluating these means of measurements may be important for future studies investigating the effect of PROSE wear on intraocular pressure.

DETAILED DESCRIPTION:
The goal of this research is to determine the reproducibility of measurements of intraocular pressure (IOP) when a scleral lens is on the eye.

This is a prospective study of the reproducibility of three non-traditional means of IOP measurements: scleral tonopen, scleral pneumatonometry, and transpalpebral Diaton tonometer. Evaluating these means of measurements may be important for future studies investigating the effect of PROSE wear on intraocular pressure.

Inclusion and Exclusion Criteria

The participant will be eligible to participate if the following criteria apply:

1. Written Informed Consent has been obtained prior to any study-related procedures taking place
2. Written documentation has been obtained in accordance with the relevant county and local privacy requirements, where applicable
3. Male or female, 18 years of age and older prior to the initial visit
4. Is an established wearer of PROSE in both eyes; without fenestrations or channels; with diameter equal to or greater than 18.0 mm
5. Upon examination by the investigator, there is adequate exposure of the sclera as required for IOP measurements with the planned device
6. In the opinion of the investigator, the subject has the ability to follow study instructions
7. In the opinion of the investigator, the subject has the ability to complete all study procedures and visits

The participant would not be eligible to participate if at least one of the following criteria is met:

1. Is aphakic (i.e., missing their natural lens inside the eye)
2. Is currently participating in any other type of eye-related clinical or research study
3. Is pregnant or nursing as reported by the subject
4. Less than 18 years of age
5. Has a condition or is in a situation which, in the investigator's opinion, may put the subject at significant risk, may confound study outcomes, or may significantly interfere with the subject's participation in the study
6. Has had previous ocular surgery within the past 12 weeks
7. Has a diagnosis of glaucoma, glaucoma suspect, ocular hypertension or prior glaucoma surgery

The following special populations will be excluded from this study:

* Adults unable to consent (including adults unable to read and understand English)
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Employees of BostonSight

Vulnerable Populations

The following special populations will be excluded from this study:

* Adults unable to consent (including adults unable to read and understand English)
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Employees of BostonSight

Number of Subjects A minimum of 30 subjects will be enrolled in this study with 10 subjects in each of the three cohorts. This is a low risk study. The investigators can expect an approximate 10% drop-out rate, so the investigators will expect to recruit approximately 33 subjects; and the first 30 to be eligible and complete the study will be used for data analysis.

The first 10 subjects will be randomly chosen for the first cohort (scleral TonoPen), the second 10 subjects will be randomly chosen for the second cohort (scleral pneumatonometry), and the third 10 subjects will be randomly chosen for the third cohort (Diaton).

Recruitment Methods Recruitment will begin once IRB approval has been received and will occur through BostonSight. The subject pool will consist of patients who are actively coming through the clinic. The investigators anticipate that all our subjects will be from the current patient population at BostonSight. Patients will be recruited via mailing and/or email and at office visits. If a patient is interested in participating in the study, they will be directed to the principal investigator or the study coordinator who will go over the study and ask the screening questions. If they are eligible based on the screening criteria, they will be invited for participation in the study. If the person calls to learn about the study, the investigator or coordinator will use the outline to determine initial eligibility. Current patients of BostonSight may also be recruited as a result of a search of the patient database. A partial HIPAA waiver is requested to permit the investigators to use the database to identify prospective patients.

The primary endpoints in this study are as follows:

1. Intraocular pressure

1. Tonopen, scleral with PD
2. Pneumatonometer, scleral with PD
3. Diaton, transpalpebral with PD

Procedures Involved Once a subject has been identified, the initial visit will be scheduled.

During the visit:

1. Informed consent will be completed
2. Record the patient's general medical history and habitual contact lens information, including lens design, power, and diameter.
3. An investigator will conduct visual acuity assessments of both eyes (Snellen).
4. Assess the fit of the PROSE device via slit lamp assessment of both eyes.
5. Assess the cornea and conjunctiva of both eyes with the PROSE device on and off.
6. The investigator will instill one drop of topical anesthetic in both eyes followed by a lubricating preservative-free artificial tear drop, such as Refresh Plus, prior to IOP measurements.
7. Measure intraocular pressure of both eyes with the PD on via (method depends on which cohort subject is in):

   1. Scleral TonoPen
   2. Scleral pneumatonometry
   3. Transpalpebral Diaton
8. Assess the conjunctiva of both eyes after measurement with the PD on

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent has been obtained prior to any study-related procedures taking place
2. Written documentation has been obtained in accordance with the relevant county and local privacy requirements, where applicable
3. Male or female, 18 years of age and older prior to the initial visit
4. Is an established wearer of PROSE in both eyes; without fenestrations or channels; with diameter equal to or greater than 18.0 mm
5. Upon examination by the investigator, there is adequate exposure of the sclera as required for IOP measurements with the planned device
6. In the opinion of the investigator, the subject has the ability to follow study instructions
7. In the opinion of the investigator, the subject has the ability to complete all study procedures and visits

Exclusion Criteria:

1. Is aphakic (i.e., missing their natural lens inside the eye)
2. Is currently participating in any other type of eye-related clinical or research study
3. Is pregnant or nursing as reported by the subject
4. Less than 18 years of age
5. Has a condition or is in a situation which, in the investigator's opinion, may put the subject at significant risk, may confound study outcomes, or may significantly interfere with the subject's participation in the study
6. Has had previous ocular surgery within the past 12 weeks
7. Has a diagnosis of glaucoma, glaucoma suspect, ocular hypertension or prior glaucoma surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Brocks, MD, Principal Investigator — Boston Sight
Locations (1):
- BostonSight, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We do not anticipate the need to share but will publish findings

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Scleral Tonopen | Scleral Pneumatonometer | Diaton
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were 18 years of age or older and were recruited from a pool of current clinic patients who carried the diagnosis of corneal ectasia and were established bilateral wearers of a PD with diameters of 18.0 mm or greater and an optimized fit (as determined by their current dispensing optometrist and confirmed at the study slit-lamp examination).
Groups:
- Scleral Tonopen: IOP for this group is measured using a scleral tonopen
- Scleral Pneumatonometry: IOP for this group is measured using scleral pneumatonometry
- Diaton: IOP for this group is measured using Diaton
- Total: Total of all reporting groups
Arm/Group | Scleral Tonopen | Scleral Pneumatonometry | Diaton | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 9 | 29
  >=65 years | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.80 (10.14) | 50.80 (7.74) | 46.77 (10.82) | 47.33 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 4 | 14
  Male | 3 | 7 | 6 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30
mean IOP [Mean (Standard Deviation); unit: mmHg] | 24.23 (8.59) | 22.32 (6.41) | 24.52 (12.20) | 23.275 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: The Goal of This Research is to Determine the Reproducibility of Measurements of Intraocular Pressure (IOP) When a Scleral Lens is on the Eye.
Description: Intraocular pressure will be measured using one of three different tonometers. The reproducibility of measurements on each device will be studied.
Time Frame: patient will participate for 1 hour
Population: Participants were 18 years of age or older and were recruited from a pool of current clinic patients who carried the diagnosis of corneal ectasia and were established bilateral wearers of a PROSE device.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Tonopen: IOP reproducibility evaluated using Tonopen
- Scleral Pneumotonometry: IOP reproducibility evaluated using Pneumatonometry
- Diaton: IOP reproducibility evaluated using Diaton
Arm/Group | Tonopen | Scleral Pneumotonometry | Diaton
Number analyzed (Participants) | 10 | 10 | 10
mmHg | 24.23 (8.59) | 22.32 (6.41) | 24.52 (12.20)
Statistical Analysis 1: Comparison: Tonopen vs Scleral Pneumotonometry; Test type: Other — The mean and standard deviation was analyzed; p = 0.07, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 day
Description: All patients were monitored for adverse events or serious adverse events.
Groups:
- Scleral Tonopen: Intraocular pressure for this group is measured using a scleral tonopen
- Scleral Pneumatonometry: Intraocular pressure for this group is measured using a scleral pneumatonometry
- Diaton: Intraocular pressure for this group is measured using a Diaton
Arm/Group | Scleral Tonopen | Scleral Pneumatonometry | Diaton
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT04308941/Prot_002.pdf
  • Informed Consent Form (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT04308941/ICF_006.pdf